CLINICAL TRIAL: NCT05504252
Title: METIMMOX-2: Metastatic pMMR/MSS Colorectal Cancer - Shaping Anti-Tumor Immunity by Oxaliplatin
Acronym: METIMMOX-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Prof Dr Anne Hansen Ree, Principal Investigator, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-500027-76-00; 2022-500027-76-00 (Other: European Medicines Agency (CTIS))
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Adenocarcinoma; Mucinous Adenocarcinoma; Signet Ring Cell Adenocarcinoma
Keywords: Immune checkpoint inhibitor (nivolumab); Oxaliplatin
MeSH Terms: conditions — Adenocarcinoma, Mucinous; Carcinoma, Signet Ring Cell | interventions — Nivolumab; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Arm (Experimental): The study has a start-up single-arm design consisting of 2 cycles of the Nordic FLOX regimen followed by 2 cycles of nivolumab for a total of 4 individual cycles before radiologic response assessment and patient stratification to continued therapy or not.
  Patients who present less than 10% target lesion reduction at the first radiologic response assessment will proceed to standard-of-care treatment at the Clinical Investigator's discretion.
  Patients who present 10% or higher target lesion reduction at the first radiologic response assessment will continue with alternating 2 cycles of the Nordic FLOX regimen and 2 cycles of nivolumab in a go-and-stop schedule until progressive disease on ongoing therapy (defining PFS), intolerable toxicity, withdrawal of consent, or death, whichever occurs first.
  Interventions: Drug: Nivolumab; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Nivolumab — Q2W
  Nivolumab: 240 mg fixed dose over 30 minutes, IV administration every 2 weeks
  Other Names: Opdivo
Drug: Oxaliplatin — FLOX, Q2W
  Other Names: 5-fluorouracil; folinic acid

SUMMARY:
Hypothesis: Patients with metastatic colorectal cancer with DNA mismatch repair-proficient (pMMR) function / microsatellite-stable (MSS) phenotype harbor a non-immunogenic disease that can be transformed into an immunogenic condition by short-course oxaliplatin-based therapy, and may achieve durable disease control or even tumor eradication by the addition of immune checkpoint blockade therapy to the standard-of-care oxaliplatin-based treatment.

DETAILED DESCRIPTION:
The study has a start-up single-arm design consisting of 2 cycles of the Nordic FLOX regimen followed by 2 cycles of nivolumab for a total of 4 individual cycles (8 weeks, or longer if cycles have been delayed) before radiologic response assessment and patient stratification to continued therapy.

Patients who present less than 10% target lesion reduction at the first radiologic response assessment will proceed to standard-of-care treatment at the Clinical Investigator's discretion. Patients will be followed for PFS (from the date of study enrolment).

Patients who present 10% or higher target lesion reduction at the first radiologic response assessment will continue treatment with alternating 2 cycles of the Nordic FLOX regimen and 2 cycles of nivolumab. From the time of stratification, radiologic response assessment will be every 8 weeks. After a total of 12 individual cycles (4 initial cycles followed by 8 continuation cycles; Sequence 1), patients will enter a break that will persist until disease progression, following radiologic assessment every 8 weeks during the break, when therapy is reintroduced and administered for another total of 12 individual cycles (Sequence 2) before a new break. This go-and-stop schedule will be continued until progressive disease on ongoing therapy (defining PFS), intolerable toxicity, withdrawal of consent, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically verified pMMR/MSS colorectal adenocarcinoma (also comprising the mucinous adenocarcinoma and signet-ring cell carcinoma entities).
* Patient is ambulatory with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patient is at least 18 years of age.
* Patient has radiologically measurable metastatic disease.
* Patient has an infradiaphragmatic metastatic lesion that can be biopsied.
* Patient has not had previous systemic cytotoxic therapy for the metastatic disease, except for previous neoadjuvant treatment.
* Patient is eligible for the Nordic FLOX regimen when it would be the preferred treatment option for first-line therapy in routine practice.
* Patient has the following laboratory values, as measured in serum/plasma within 14 days prior to study entry, indicative of adequate organ function:

  * Hemoglobin at least 10.0 g/dL
  * Neutrophils at least 1.5 x10(9)/L (without current use of colony-stimulating factors).
  * Platelets at least 100 x10(9)/L. - C-reactive protein less than 60 mg/L
  * AST/ALT no higher than 2xULN when patient does not have metastatic disease in the liver or no higher than 5xULN when patient has metastatic disease in the liver. o Bilirubin no higher than 1.5xULN when patient does not have metastatic disease in the liver or no higher than 2xULN when patient has metastatic disease in the liver
  * Albumin no lower than 30 g/L. - INR within normal level
  * Creatinine no higher than 1.5xULN
* Woman of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
* WOCBP will use an adequate method to avoid pregnancy for a period of 26 weeks (which includes the required 30 days plus the time required for nivolumab to undergo five half-lives) after the last therapy dose
* Woman is not breastfeeding
* Male who is sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 26 weeks (which includes the required time to ensure duration of sperm turnover plus the time required for the investigational drugs to undergo five half-lives) after the last therapy dose
* Signed informed consent form and expected cooperation of the patients for the treatment and follow-up must be obtained and documented according to International Conference on Harmonization - Good Clinical Practice and national/local regulations

Exclusion Criteria:

* Patient has metastatic dMMR/MSI colorectal cancer.
* Patient has initially resectable metastatic disease for which neoadjuvant therapy is deemed superfluous.
* Patient has supradiaphragmatic metastatic disease as the sole site(s).
* Patient has untreated or symptomatic brain metastasis (patient must be symptom-free without the use of corticosteroids).
* Patient has experienced a period of less than 6 months since discontinuation of neoadjuvant or adjuvant oxaliplatincontaining chemotherapy.
* Patient is ineligible for full (100%) chemotherapy doses at first treatment cycle.
* Patient has partial or complete dihydropyrimidine dehydrogenase (DPD) deficiency.
* Patient has had radiation therapy against the only measurable lesion within 4 weeks of start of study treatment.
* Patient has a medical condition treated with anticoagulant medication that cannot be replaced by low molecular weight heparin or a direct oral anticoagulant during active study treatment.
* Patient has a nervous system disorder worse than CTCAE grade 1.
* Patient has any medical condition that will preclude him/her from immune checkpoint blockade therapy, such as:

  * Active or chronic hepatitis B or hepatitis C. - Known history of human immunodeficiency virus or acquired immunodeficiency-related illnesses.
  * Diagnosis of immunodeficiency or medical condition requiring systemic steroids or other forms of immunosuppressive therapy.
  * Autoimmune disease that has required systemic therapy within the past 2 years.
  * Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study therapy.
  * Active infection or chronic infection requiring chronic suppressive antibiotics.
  * Known history of previous diagnosis of tuberculosis.
* Patient with current or prior use of immunosuppressive medication within 28 days before the first dose of study therapy, with the exceptions of intranasal corticosteroids or systemic corticosteroids at physiological doses that do not exceed 10mg/day of prednisone or an equivalent corticosteroid.
* Patient has any medical condition or needs to use medication, as listed in the SmPC of each Investigational Medical Product (IMP), that will preclude him/her from receiving treatment with IMP, such as:

  * Pernicious anemia or anemias due to vitamin B12 deficiency (SmPC-listed contraindications for folinic acid).
  * A known complete absence of DPD activity.
  * Has been treated with brivudine, sorivudine, or their chemically related analogs, which are potent inhibitors of the enzyme DPD that degrades fluorouracil. Fluorouracil must not be taken within 4 weeks of treatment with brivudine, sorivudine, or their chemically related analogs.
  * Other SmPC-listed contraindications for the IMPs are covered by other exclusion criteria.
* Patient has undergone treatment with any IMP that may interfere with the study treatment within 4 weeks prior to first administration of study drug.
* Patient has known hypersensitivity to any of the study IMP components.
* Patient has history of other prior malignancy, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin, cervical cancer stage IB, stage I prostate cancer considered not necessary to treat, and another malignancy that was treated with curative intent more than 5 years ago and has not relapsed later.
* Patient has significant cardiac, pulmonary, or other medical illness that would limit activity of daily life or survival.
* Patient is pregnant or breastfeeding.
* Patient has any other reason, in the opinion of Clinical Investigator, not to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of the first FLOX cycle until the date of disease progression on ongoing therapy or death, whichever occurs first, assessed up to 60 months
  To determine PFS, in terms of continuation of treatment strategy, of repeat sequential treatment with the Nordic FLOX regimen and nivolumab in patients with previously untreated unresectable metastatic pMMR/MSS colorectal cancer reaching 10% or higher target lesion reduction at the first radiologic restaging.

SECONDARY OUTCOMES:
Incidence of adverse events | From date of the first FLOX cycle until 100 days following discontinuation of the study treatment, assessed up to 60 months
  Safety
Grading of adverse events | From date of the first FLOX cycle until 100 days following discontinuation of the study treatment, assessed up to 60 months
  Tolerability
Objective response rate | Through study completion, an average of 18 months
  ORR
Duration of response | From date of the best overall response until the date of disease progression, assessed up to 60 months
  DoR
Secondary surgical curative-intent resection rate | Through study completion, an average of 18 months
  SSCiR
Overall survival | From date of the first FLOX cycle until the date of death, assessed up to 60 months
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Christian Kersten, MD, PhD, Study Chair — University Hospital, Akershus
Locations (3):
- Norway (3):
  - Akershus University Hospital, Lørenskog, Akershus
  - Oslo University Hospital, Oslo, Akershus
  - St Olavs Hospital, Trondheim, Trøndelag

IPD SHARING:
Plan to Share IPD: Yes
The listed study information can be made available from the Principal Investigator on reasonable request and in accordance with the General Data Protection Regulation of the European Union.
Supporting Information: Study Protocol, CSR
Time Frame: 2022-2047
Access Criteria: The listed study information can be made available from the Principal Investigator on reasonable request and in accordance with the General Data Protection Regulation of the European Union.

REFERENCES:
- [Background] Abrahamsson H, Jensen BV, Berven LL, Nielsen DL, Saltyte Benth J, Johansen JS, Larsen FO, Johansen JS, Ree AH. Antitumour immunity invoked by hepatic arterial infusion of first-line oxaliplatin predicts durable colorectal cancer control after liver metastasis ablation: 8-12 years of follow-up. Int J Cancer. 2020 Apr 1;146(7):2019-2026. doi: 10.1002/ijc.32847. Epub 2020 Jan 7. PMID 31872440
- [Background] Andre T, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Bendell J, Le DT, Yoshino T, Van Cutsem E, Yang P, Farooqui MZH, Marinello P, Diaz LA Jr; KEYNOTE-177 Investigators. Pembrolizumab in Microsatellite-Instability-High Advanced Colorectal Cancer. N Engl J Med. 2020 Dec 3;383(23):2207-2218. doi: 10.1056/NEJMoa2017699. PMID 33264544
- [Background] Bains SJ, Abrahamsson H, Flatmark K, Dueland S, Hole KH, Seierstad T, Redalen KR, Meltzer S, Ree AH. Immunogenic cell death by neoadjuvant oxaliplatin and radiation protects against metastatic failure in high-risk rectal cancer. Cancer Immunol Immunother. 2020 Mar;69(3):355-364. doi: 10.1007/s00262-019-02458-x. Epub 2019 Dec 31. PMID 31893287
- [Background] Borcoman E, Kanjanapan Y, Champiat S, Kato S, Servois V, Kurzrock R, Goel S, Bedard P, Le Tourneau C. Novel patterns of response under immunotherapy. Ann Oncol. 2019 Mar 1;30(3):385-396. doi: 10.1093/annonc/mdz003. PMID 30657859
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Dagenborg VJ, Marshall SE, Yaqub S, Grzyb K, Boye K, Lund-Iversen M, Hoye E, Berstad AE, Fretland AA, Edwin B, Ree AH, Flatmark K. Neoadjuvant chemotherapy is associated with a transient increase of intratumoral T-cell density in microsatellite stable colorectal liver metastases. Cancer Biol Ther. 2020 May 3;21(5):432-440. doi: 10.1080/15384047.2020.1721252. Epub 2020 Feb 26. PMID 32098573
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Galluzzi L, Vitale I, Warren S, Adjemian S, Agostinis P, Martinez AB, Chan TA, Coukos G, Demaria S, Deutsch E, Draganov D, Edelson RL, Formenti SC, Fucikova J, Gabriele L, Gaipl US, Gameiro SR, Garg AD, Golden E, Han J, Harrington KJ, Hemminki A, Hodge JW, Hossain DMS, Illidge T, Karin M, Kaufman HL, Kepp O, Kroemer G, Lasarte JJ, Loi S, Lotze MT, Manic G, Merghoub T, Melcher AA, Mossman KL, Prosper F, Rekdal O, Rescigno M, Riganti C, Sistigu A, Smyth MJ, Spisek R, Stagg J, Strauss BE, Tang D, Tatsuno K, van Gool SW, Vandenabeele P, Yamazaki T, Zamarin D, Zitvogel L, Cesano A, Marincola FM. Consensus guidelines for the definition, detection and interpretation of immunogenic cell death. J Immunother Cancer. 2020 Mar;8(1):e000337. doi: 10.1136/jitc-2019-000337. PMID 32209603
- [Background] Grasso CS, Giannakis M, Wells DK, Hamada T, Mu XJ, Quist M, Nowak JA, Nishihara R, Qian ZR, Inamura K, Morikawa T, Nosho K, Abril-Rodriguez G, Connolly C, Escuin-Ordinas H, Geybels MS, Grady WM, Hsu L, Hu-Lieskovan S, Huyghe JR, Kim YJ, Krystofinski P, Leiserson MDM, Montoya DJ, Nadel BB, Pellegrini M, Pritchard CC, Puig-Saus C, Quist EH, Raphael BJ, Salipante SJ, Shin DS, Shinbrot E, Shirts B, Shukla S, Stanford JL, Sun W, Tsoi J, Upfill-Brown A, Wheeler DA, Wu CJ, Yu M, Zaidi SH, Zaretsky JM, Gabriel SB, Lander ES, Garraway LA, Hudson TJ, Fuchs CS, Ribas A, Ogino S, Peters U. Genetic Mechanisms of Immune Evasion in Colorectal Cancer. Cancer Discov. 2018 Jun;8(6):730-749. doi: 10.1158/2159-8290.CD-17-1327. Epub 2018 Mar 6. PMID 29510987
- [Background] Guinney J, Dienstmann R, Wang X, de Reynies A, Schlicker A, Soneson C, Marisa L, Roepman P, Nyamundanda G, Angelino P, Bot BM, Morris JS, Simon IM, Gerster S, Fessler E, De Sousa E Melo F, Missiaglia E, Ramay H, Barras D, Homicsko K, Maru D, Manyam GC, Broom B, Boige V, Perez-Villamil B, Laderas T, Salazar R, Gray JW, Hanahan D, Tabernero J, Bernards R, Friend SH, Laurent-Puig P, Medema JP, Sadanandam A, Wessels L, Delorenzi M, Kopetz S, Vermeulen L, Tejpar S. The consensus molecular subtypes of colorectal cancer. Nat Med. 2015 Nov;21(11):1350-6. doi: 10.1038/nm.3967. Epub 2015 Oct 12. PMID 26457759
- [Background] Hadden WJ, de Reuver PR, Brown K, Mittal A, Samra JS, Hugh TJ. Resection of colorectal liver metastases and extra-hepatic disease: a systematic review and proportional meta-analysis of survival outcomes. HPB (Oxford). 2016 Mar;18(3):209-20. doi: 10.1016/j.hpb.2015.12.004. Epub 2016 Feb 1. PMID 27017160
- [Background] Hoos A, Wolchok JD, Humphrey RW, Hodi FS. CCR 20th Anniversary Commentary: Immune-Related Response Criteria--Capturing Clinical Activity in Immuno-Oncology. Clin Cancer Res. 2015 Nov 15;21(22):4989-91. doi: 10.1158/1078-0432.CCR-14-3128. PMID 26567357
- [Background] Kalanxhi E, Meltzer S, Schou JV, Larsen FO, Dueland S, Flatmark K, Jensen BV, Hole KH, Seierstad T, Redalen KR, Nielsen DL, Ree AH. Systemic immune response induced by oxaliplatin-based neoadjuvant therapy favours survival without metastatic progression in high-risk rectal cancer. Br J Cancer. 2018 May;118(10):1322-1328. doi: 10.1038/s41416-018-0085-y. Epub 2018 Apr 26. PMID 29695770
- [Background] Lee JW, Stone ML, Porrett PM, Thomas SK, Komar CA, Li JH, Delman D, Graham K, Gladney WL, Hua X, Black TA, Chien AL, Majmundar KS, Thompson JC, Yee SS, O'Hara MH, Aggarwal C, Xin D, Shaked A, Gao M, Liu D, Borad MJ, Ramanathan RK, Carpenter EL, Ji A, de Beer MC, de Beer FC, Webb NR, Beatty GL. Hepatocytes direct the formation of a pro-metastatic niche in the liver. Nature. 2019 Mar;567(7747):249-252. doi: 10.1038/s41586-019-1004-y. Epub 2019 Mar 6. PMID 30842658
- [Background] Lenz HJ, Van Cutsem E, Luisa Limon M, Wong KYM, Hendlisz A, Aglietta M, Garcia-Alfonso P, Neyns B, Luppi G, Cardin DB, Dragovich T, Shah U, Abdullaev S, Gricar J, Ledeine JM, Overman MJ, Lonardi S. First-Line Nivolumab Plus Low-Dose Ipilimumab for Microsatellite Instability-High/Mismatch Repair-Deficient Metastatic Colorectal Cancer: The Phase II CheckMate 142 Study. J Clin Oncol. 2022 Jan 10;40(2):161-170. doi: 10.1200/JCO.21.01015. Epub 2021 Oct 12. PMID 34637336
- [Background] Liao W, Overman MJ, Boutin AT, Shang X, Zhao D, Dey P, Li J, Wang G, Lan Z, Li J, Tang M, Jiang S, Ma X, Chen P, Katkhuda R, Korphaisarn K, Chakravarti D, Chang A, Spring DJ, Chang Q, Zhang J, Maru DM, Maeda DY, Zebala JA, Kopetz S, Wang YA, DePinho RA. KRAS-IRF2 Axis Drives Immune Suppression and Immune Therapy Resistance in Colorectal Cancer. Cancer Cell. 2019 Apr 15;35(4):559-572.e7. doi: 10.1016/j.ccell.2019.02.008. Epub 2019 Mar 21. PMID 30905761
- [Background] Meltzer S, Torgunrud A, Abrahamsson H, Solbakken AM, Flatmark K, Dueland S, Bakke KM, Bousquet PA, Negard A, Johansen C, Lyckander LG, Larsen FO, Schou JV, Redalen KR, Ree AH. The circulating soluble form of the CD40 costimulatory immune checkpoint receptor and liver metastasis risk in rectal cancer. Br J Cancer. 2021 Jul;125(2):240-246. doi: 10.1038/s41416-021-01377-y. Epub 2021 Apr 9. PMID 33837301
- [Background] Overman MJ, McDermott R, Leach JL, Lonardi S, Lenz HJ, Morse MA, Desai J, Hill A, Axelson M, Moss RA, Goldberg MV, Cao ZA, Ledeine JM, Maglinte GA, Kopetz S, Andre T. Nivolumab in patients with metastatic DNA mismatch repair-deficient or microsatellite instability-high colorectal cancer (CheckMate 142): an open-label, multicentre, phase 2 study. Lancet Oncol. 2017 Sep;18(9):1182-1191. doi: 10.1016/S1470-2045(17)30422-9. Epub 2017 Jul 19. PMID 28734759
- [Background] Pfirschke C, Engblom C, Rickelt S, Cortez-Retamozo V, Garris C, Pucci F, Yamazaki T, Poirier-Colame V, Newton A, Redouane Y, Lin YJ, Wojtkiewicz G, Iwamoto Y, Mino-Kenudson M, Huynh TG, Hynes RO, Freeman GJ, Kroemer G, Zitvogel L, Weissleder R, Pittet MJ. Immunogenic Chemotherapy Sensitizes Tumors to Checkpoint Blockade Therapy. Immunity. 2016 Feb 16;44(2):343-54. doi: 10.1016/j.immuni.2015.11.024. Epub 2016 Feb 9. PMID 26872698
- [Background] Rahma OE, Hodi FS. The Intersection between Tumor Angiogenesis and Immune Suppression. Clin Cancer Res. 2019 Sep 15;25(18):5449-5457. doi: 10.1158/1078-0432.CCR-18-1543. Epub 2019 Apr 3. PMID 30944124
- [Background] Ree AH, Nygaard V, Russnes HG, Heinrich D, Nygaard V, Johansen C, Bergheim IR, Hovig E, Beiske K, Negard A, Borresen-Dale AL, Flatmark K, Maelandsmo GM. Responsiveness to PD-1 Blockade in End-Stage Colon Cancer with Gene Locus 9p24.1 Copy-Number Gain. Cancer Immunol Res. 2019 May;7(5):701-706. doi: 10.1158/2326-6066.CIR-18-0777. Epub 2019 Feb 25. PMID 30804006
- [Background] Smyth MJ, Ngiow SF, Ribas A, Teng MW. Combination cancer immunotherapies tailored to the tumour microenvironment. Nat Rev Clin Oncol. 2016 Mar;13(3):143-58. doi: 10.1038/nrclinonc.2015.209. Epub 2015 Nov 24. PMID 26598942
- [Background] Stremitzer S, Vermeulen P, Graver S, Kockx M, Dirix L, Yang D, Zhang W, Stift J, Wrba F, Gruenberger T, Lenz HJ, Scherer SJ. Immune phenotype and histopathological growth pattern in patients with colorectal liver metastases. Br J Cancer. 2020 May;122(10):1518-1524. doi: 10.1038/s41416-020-0812-z. Epub 2020 Mar 24. PMID 32205863
- [Background] Sveen A, Kopetz S, Lothe RA. Biomarker-guided therapy for colorectal cancer: strength in complexity. Nat Rev Clin Oncol. 2020 Jan;17(1):11-32. doi: 10.1038/s41571-019-0241-1. Epub 2019 Jul 9. PMID 31289352
- [Background] Tesniere A, Schlemmer F, Boige V, Kepp O, Martins I, Ghiringhelli F, Aymeric L, Michaud M, Apetoh L, Barault L, Mendiboure J, Pignon JP, Jooste V, van Endert P, Ducreux M, Zitvogel L, Piard F, Kroemer G. Immunogenic death of colon cancer cells treated with oxaliplatin. Oncogene. 2010 Jan 28;29(4):482-91. doi: 10.1038/onc.2009.356. Epub 2009 Nov 2. PMID 19881547
- [Background] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Background] Whiteside TL, Demaria S, Rodriguez-Ruiz ME, Zarour HM, Melero I. Emerging Opportunities and Challenges in Cancer Immunotherapy. Clin Cancer Res. 2016 Apr 15;22(8):1845-55. doi: 10.1158/1078-0432.CCR-16-0049. PMID 27084738
- [Background] Zitvogel L, Kepp O, Senovilla L, Menger L, Chaput N, Kroemer G. Immunogenic tumor cell death for optimal anticancer therapy: the calreticulin exposure pathway. Clin Cancer Res. 2010 Jun 15;16(12):3100-4. doi: 10.1158/1078-0432.CCR-09-2891. Epub 2010 Apr 26. PMID 20421432
- [Background] Ostrup O, Dagenborg VJ, Rodland EA, Skarpeteig V, Silwal-Pandit L, Grzyb K, Berstad AE, Fretland AA, Maelandsmo GM, Borresen-Dale AL, Ree AH, Edwin B, Nygaard V, Flatmark K. Molecular signatures reflecting microenvironmental metabolism and chemotherapy-induced immunogenic cell death in colorectal liver metastases. Oncotarget. 2017 Jul 18;8(44):76290-76304. doi: 10.18632/oncotarget.19350. eCollection 2017 Sep 29. PMID 29100312